CLINICAL TRIAL: NCT02800460
Title: Development of New Multi-contrasts Approaches by Magnetic Resonance Imaging at 3 Tesla Dedicated to Targeting Subthalamic Nucleus on Parkinsonian Patients.
Brief Title: New Approaches in MRI at 3T Dedicated to Targeting Subthalamic Nucleus on Parkinsonian Patients
Acronym: Optimise_3T
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: C15-90; 2016-A00231-50 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-06-01; First posted 2016-06-15 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Subthalamic nucleus; Basal ganglia; Parkinson disease; Magnetic Resonance Imaging; Susceptibility-Weighted Imaging
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Deep brain stimulation with fMRI-3T (Other): Patients will have a 3T-fMRI before their usual MRI-1,5T
  Interventions: Procedure: fMRI-3T

INTERVENTIONS:
Procedure: fMRI-3T — fMRI-3T will be performed during the visit 1: day of anesthesia consultation (this fMRI-3T will last approximately one hour)

SUMMARY:
Deep brain stimulation (DBS) of the subthalamic nucleus (STN) is a validated procedure, used in many French and international centers for the treatment of severe forms of Parkinson's disease (PD). The improvement of parkinsonian motor symptoms by stimulation of the STN is 50 to 80% on average. The main advantage of DBS is that the surgery has low morbidity and mortality, it is adaptable to the patient's symptoms and its effect is reversible. This treatment is now a routine and more than 85,000 patients worldwide have benefited from the installation of this system. Since 1997, this treatment is available to patients followed in the Pitié Salpêtrière (GHPS).

The accuracy of preoperative anatomic targeting in stereotactic neurosurgery will improve with the use of high-field MRI. However, several new issues and inherent in that high-field MRI should be evaluated before the images can be used directly.

The chosen sequences must be short to be feasible, minimizing patient discomfort, and evaluated on several patients to ensure the low interindividual variability. In addition, the quality of the display on all of the sections should provide a reliable three-dimensional information. Finally, the quality of targeting and its possible improvement should be checked.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of the subthalamic nucleus (STN) is a validated procedure, used in many French and international centers for the treatment of severe forms of Parkinson's disease (PD). The improvement of parkinsonian motor symptoms by stimulation of the STN is 50 to 80% on average. The main advantage of DBS is that the surgery has low morbidity and mortality, it is adaptable to the patient's symptoms and that its effect is reversible. This treatment is now a routine and more than 85,000 patients worldwide have benefited from the installation of this system. Since 1997, this treatment is available to patients followed in the Pitié Salpêtrière (GHPS).

The quality of the implantation of stimulating electrodes into deep brain structures to achieve, particularly in the NST for PD patients, is crucial to obtain an excellent result. Accurate identification of these deep nuclei and especially the NST on MRI of each patient to be operated is an essential step and directly affects the smooth running of the surgery and the final clinical outcome.

The visualization of the NST on MRI remains difficult, variable between patients, requiring specific sequences or even sequences dedicated to this activity. In GHPS the investigators opted for the realization of an efficient particular sequence for viewing the NST but the latter has several disadvantages the first being its duration. Indeed, the patient needs to keep still, head fixed for 40 minutes, and this major constraint is sometimes impossible due to the importance of abnormal movements. The second is the variability between patients with visualization being sometimes inconspicuous. The third is the susceptibility of this sequence to flow artifacts at the level of the third ventricle that significantly disrupt viewing NST.

The new MRI techniques available for some years, especially at 3 Tesla should allow better visualization of the deep nuclei of the brain and NST in particular. Indeed, the high-field MRI has become an indispensable tool for both define the morphological and structural features but also functional and metabolic deep nuclei of the brain, particularly the NST.

The accuracy of preoperative anatomic targeting in stereotactic neurosurgery will improve with the use of high-field MRI. However, several new issues and inherent in that high-field MRI should be evaluated before the images can be used directly.

The chosen sequence must be short to be feasible, minimizing patient discomfort, and evaluated several patients to ensure the low interindividual variability. In addition, the quality of the display on all of the sections should provide a reliable three-dimensional information. Finally, the quality of targeting and its possible improvement should be checked.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease (according to the criteria of the "United Kingdom Parkinson's Disease Society Brain Bank";
* Age between 18 and 70 years
* motor complications in the form of fluctuations in motor state or induced dyskinesias dopaminergic therapy, despite optimal medical treatment;
* Excellent responsiveness to levodopa (improved motor UPDRS score of higher than 50% during the acute test with levodopa)
* People who voluntarily accepted and intelligently participate in the study (signing a written consent)
* Patient receiving social health insurance

Exclusion Criteria:

* Patients carry an apomorphine pump used in single and continuous treatment;
* scalable psychiatric pathology;
* Dementia (MMS <24/30);
* Existence of against-indications to MRI (cardiac or neural stimulator, ferromagnetic surgical clips, implants and metal objects, intraocular foreign bodies, pregnancy, claustrophobia).
* Persons under guardianship, trusteeship or any other administrative or judicial deprivation of rights and freedom

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2025-06-08 (Actual); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Measure of the distance between two target points within the NST defined on a optimized Flair sequence on a research 3T MRI and on a routine T2 sequence acquired at 1.5T. | Visit 3 : day of surgery
  The measure will be performed with the new 3T MRI (Flair sequence) conducted as part of this protocol and the clinical routine on the 1,5T MRI (T2 sequences).

SECONDARY OUTCOMES:
Measure of target contouring with a quantitative scale | Visit 3: Day of surgery
  Target contouring from 3T-fMRI and from 1,5T-MRI
Measure of target volume | Visit 3: Day of surgery
  Volume measures with 3T-fMRI and with the 1.5-MRI

CONTACTS AND LOCATIONS:
Locations (1):
- GHPS, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benabid AL, Koudsie A, Benazzouz A, Piallat B, Krack P, Limousin-Dowsey P, Lebas JF, Pollak P. Deep brain stimulation for Parkinson's disease. Adv Neurol. 2001;86:405-12. No abstract available. PMID 11554003
- [Background] Bejjani BP, Dormont D, Pidoux B, Yelnik J, Damier P, Arnulf I, Bonnet AM, Marsault C, Agid Y, Philippon J, Cornu P. Bilateral subthalamic stimulation for Parkinson's disease by using three-dimensional stereotactic magnetic resonance imaging and electrophysiological guidance. J Neurosurg. 2000 Apr;92(4):615-25. doi: 10.3171/jns.2000.92.4.0615. PMID 10761650
- [Background] Egidi M, Rampini P, Locatelli M, Farabola M, Priori A, Pesenti A, Tamma F, Caputo E, Chiesa V, Villani RM. Visualisation of the subthalamic nucleus: a multiple sequential image fusion (MuSIF) technique for direct stereotaxic localisation and postoperative control. Neurol Sci. 2002 Sep;23 Suppl 2:S71-2. doi: 10.1007/s100720200075. PMID 12548349
- [Background] Longhi M, Ricciardi G, Tommasi G, Nicolato A, Foroni R, Bertolasi L, Beltramello A, Moretto G, Tinazzi M, Gerosa M. The Role of 3T Magnetic Resonance Imaging for Targeting the Human Subthalamic Nucleus in Deep Brain Stimulation for Parkinson Disease. J Neurol Surg A Cent Eur Neurosurg. 2015 May;76(3):181-9. doi: 10.1055/s-0033-1354749. Epub 2015 Mar 12. PMID 25764475
- [Background] Lefranc M, Derrey S, Merle P, Tir M, Constans JM, Montpellier D, Macron JM, Le Gars D, Peltier J, Baledentt O, Krystkowiak P. High-resolution 3-dimensional T2*-weighted angiography (HR 3-D SWAN): an optimized 3-T magnetic resonance imaging sequence for targeting the subthalamic nucleus. Neurosurgery. 2014 Jun;74(6):615-26; discussion 627. doi: 10.1227/NEU.0000000000000319. PMID 24535261
- [Background] Yelnik J, Bardinet E, Dormont D, Malandain G, Ourselin S, Tande D, Karachi C, Ayache N, Cornu P, Agid Y. A three-dimensional, histological and deformable atlas of the human basal ganglia. I. Atlas construction based on immunohistochemical and MRI data. Neuroimage. 2007 Jan 15;34(2):618-38. doi: 10.1016/j.neuroimage.2006.09.026. Epub 2006 Nov 15. PMID 17110133
- [Background] Breit S, LeBas JF, Koudsie A, Schulz J, Benazzouz A, Pollak P, Benabid AL. Pretargeting for the implantation of stimulation electrodes into the subthalamic nucleus: a comparative study of magnetic resonance imaging and ventriculography. Neurosurgery. 2006 Feb;58(1 Suppl):ONS83-95. doi: 10.1227/01.NEU.0000192689.00427.C2. PMID 16543877
- [Background] Cheng CH, Huang HM, Lin HL, Chiou SM. 1.5T versus 3T MRI for targeting subthalamic nucleus for deep brain stimulation. Br J Neurosurg. 2014 Aug;28(4):467-70. doi: 10.3109/02688697.2013.854312. Epub 2013 Nov 5. PMID 24191703
- [Background] Patil PG, Conrad EC, Aldridge JW, Chenevert TL, Chou KL. The anatomical and electrophysiological subthalamic nucleus visualized by 3-T magnetic resonance imaging. Neurosurgery. 2012 Dec;71(6):1089-95; discussion 1095. doi: 10.1227/NEU.0b013e318270611f. PMID 22948201
- [Background] Marques JP, Kober T, Krueger G, van der Zwaag W, Van de Moortele PF, Gruetter R. MP2RAGE, a self bias-field corrected sequence for improved segmentation and T1-mapping at high field. Neuroimage. 2010 Jan 15;49(2):1271-81. doi: 10.1016/j.neuroimage.2009.10.002. Epub 2009 Oct 9. PMID 19819338
- [Background] Liu T, Eskreis-Winkler S, Schweitzer AD, Chen W, Kaplitt MG, Tsiouris AJ, Wang Y. Improved subthalamic nucleus depiction with quantitative susceptibility mapping. Radiology. 2013 Oct;269(1):216-23. doi: 10.1148/radiol.13121991. Epub 2013 May 14. PMID 23674786
- [Background] Xiao Y, Fonov VS, Beriault S, Gerard I, Sadikot AF, Pike GB, Collins DL. Patch-based label fusion segmentation of brainstem structures with dual-contrast MRI for Parkinson's disease. Int J Comput Assist Radiol Surg. 2015 Jul;10(7):1029-41. doi: 10.1007/s11548-014-1119-4. Epub 2014 Sep 24. PMID 25249471
- [Background] Starr PA, Martin AJ, Ostrem JL, Talke P, Levesque N, Larson PS. Subthalamic nucleus deep brain stimulator placement using high-field interventional magnetic resonance imaging and a skull-mounted aiming device: technique and application accuracy. J Neurosurg. 2010 Mar;112(3):479-90. doi: 10.3171/2009.6.JNS081161. PMID 19681683
- [Background] Bardinet E, Belaid H, Grabli D, Welter ML, Vidal SF, Galanaud D, Derrey S, Dormont D, Cornu P, Yelnik J, Karachi C. Thalamic stimulation for tremor: can target determination be improved? Mov Disord. 2011 Feb 1;26(2):307-12. doi: 10.1002/mds.23448. Epub 2010 Dec 13. PMID 21412838